CLINICAL TRIAL: NCT07069699
Title: Phase 1b/2 Trial of Pidnarulex in MYC Aberrant Lymphoma
Brief Title: Testing the Safety of Anti-Cancer Drug, CX-5461 (Pidnarulex), in Treating Lymphoma With Specific Changes in the MYC Gene
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-04787; NCI-2025-04787 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10717 (Other: Yale University Cancer Center LAO); 10717 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2025-07-16; First posted 2025-07-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Burkitt Lymphoma; Double-Expressor Lymphoma; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Biopsy; Specimen Handling; Spinal Puncture; CX 5461; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CX-5461) (Experimental): Patients receive CX-5461 IV over 60 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo lumbar puncture with CSF collection on study and PET scan/CT scan, tumor biopsy, and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Lumbar Puncture; Drug: Pidnarulex; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo CSF and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Drug: Pidnarulex — Given IV
  Other Names: CX-5461; CX5461; Pol I Inhibitor CX5461; RNA Pol I Inhibitor CX5461
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase Ib/II trial tests the safety, side effects, best dose and how well giving CX-5461 works for the treatment of patients with B-cell non-Hodgkin lymphoma. CX-5461 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving CX-5461 may be safe, tolerable and/or effective in treating patients with B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define dose limiting toxicity (DLT). (Phase 1) II. To assess toxicity profile. (Phase 1) III. To determine the recommended phase 2 dose (RP2D). (Phase 1) IV. To perform pharmacokinetic (PK) studies. (Phase 1) V. To examine the effect of CX-5461 (Pidnarulex) on gene expression profile of MYC aberrant lymphomas. (Phase 1) VI. To determine the objective response rate (ORR) (complete response [CR] and partial response [PR]). (Phase 2)

SECONDARY OBJECTIVE:

I. To observe and record anti-tumor activity. (Phase 1 and 2)

EXPLORATORY OBJECTIVES:

I. To determine the mechanisms of response and resistance using circulating tumor deoxyribonucleic acid (ctDNA). (Phase 1 and 2) II. To observe cerebral spinal fluid (CSF) distribution of CX-5461 (Pidnarulex). (Phase 1 and 2)

OUTLINE: This is a phase 1 dose-escalation study of CX-5461 followed by a phase 2 study.

Patients receive CX-5461 intravenously (IV) over 60 minutes on days 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo lumbar puncture with cerebrospinal fluid (CSF) collection on study and positron emission tomography (PET) scan/computed tomography (CT) scan, tumor biopsy, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days, every 3-4 months for the first 2 years, and every 6 months for years 3-5.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following subtypes of aggressive B-cell non-Hodgkin lymphomas: double-expressor lymphoma (DEL), high-grade B-cell lymphoma (HGBL) with MYC and BCL2 and/or BCL6 rearrangement, or Burkitt lymphoma (BL). Eligible patients must have received at least two prior lines of treatment for diffuse large B-cell lymphoma (DLBCL) or at least one prior line of therapy for Burkitt Lymphoma and must have disease for which no standard curative or palliative treatment options exist or remain effective (Quin et al., 2016)
* Age ≥ 18 years. Because no dosing or adverse event (AE) data are currently available on the use of CX-5461 (Pidnarulex) in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%). ECOG 3 is allowed if directly related to lymphoma per treating provider
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 50,000/mcL
* Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN)

  * Patients with documented Gilbert's syndrome may be included if total bilirubin is ≤ 3 × ULN and direct bilirubin is within normal limits
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional upper limit of normal (ULN)
* Glomerular filtration rate (GFR) ≥ 60 mL/min/, calculated by multiplying the estimated (e)GFR (mL/min/1.73 m^2) by the individual's body surface area (BSA, calculated using an accepted formula) and dividing by 1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Patients with cytopenia related to abnormal bone marrow function in the setting of bone marrow involvement with lymphoma or post chimeric antigen receptor (CAR) T-cell are allowed to enroll if deemed safe by treating provider
* Patients without clinical evidence of central nervous system (CNS) lymphoma
* The effects of CX-5461 (Pidnarulex) on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) 14 days prior to study entry and for the duration of study participation and for at least 6 months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women should not breastfeed while taking CX-5461 (Pidnarulex) and for 6 months after cessation of treatment. Men treated or enrolled on this protocol must also agree to use adequate contraception 14 days prior to the study, for the duration of study participation, and 6 months after completion of CX-5461 (Pidnarulex) administration. Women of childbearing age should not donate egg(s) and men should not donate sperm for the duration of study participation and 6 months after completion of the last dose CX-5461 (Pidnarulex)
* Willingness to provide blood and biopsy samples for research purposes
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients must have recovered from clinically significant adverse events (AEs) of their most recent cancer immunotherapy to grade 1 or less (with the exception for alopecia or lymphopenia)
* Eligibility of subjects receiving any medications or substances known to affect or with the potential to affect the activity of CX-5461 (Pidnarulex) will be determined based on their potential to interact with the CYP3A4 isozyme. Specifically, subjects taking strong CYP3A4 inhibitors or strong CYP3A4 inducers will be excluded from participation in the trial. For medications or substances not listed, or in cases of uncertainty, the Principal Investigator may consult with a medical expert or a pharmacologist to make an informed decision regarding eligibility
* Patients with a baseline corrected QT (QTc) interval > 480 msec
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CX-5461 (Pidnarulex)
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because CX-5461 (Pidnarulex) is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with CX-5461 (Pidnarulex), breastfeeding should be discontinued if the mother is treated with CX-5461 (Pidnarulex)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-10-13 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (Phase 1) | Up to 30 days after last dose of study treatment
  Assessed by the Common Terminology Criteria for Adverse Events version 5. Safety will be summarized overall, by actual dose level in Phase 1b.
Recommended phase 2 dose (RP2D) (Phase 1) | Up to 5 years
Pharmacokinetic (PK) levels (Phase 1) | At cycle (C) 1 day (D) 8 at pre-dose, end of infusion, and 2 hours (hrs) post-dose; on C1D9 at 24 hrs post C1D8 infusion; on C1D10 at 48 hrs post C1D8 infusion; on C1D11 at 72 hrs post C1D8 infusion; and on C1D15 at 167 hrs post C1D8 infusion
  Assessed using Liquid Chromatography Mass Spectrometry (LC-MS).
Gene expression (Phase 1) | At baseline, C1D9 or C1D10 (within 24-48 hrs of C1D8 dosing),and at progression
  Assessed by ribonucleic acid sequencing complemented by whole exome sequencing using an average absolute log2 fold change relative to baseline with a significance threshold of p < 0.05.
Overall response rate (Phase 2) | Up to 5 years
  Assessed using standard radiographic criteria according to Lugano criteria. Phase 2 results will be reported at the RP2D.

SECONDARY OUTCOMES:
Response to therapy (Phase 1 and 2) | Up to 5 years
  Assessed according to Lugano criteria.

OTHER OUTCOMES:
Circulating tumor deoxyribonucleic acid sequencing (Phase 1 and 2) | At baseline, day 21 of cycle 1, and complete remission
PK levels of cerebrospinal fluid (Phase 1 and 2) | At C1D8 2 hours post dose
  Using LC-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Sami Ibrahimi, Principal Investigator — Yale University Cancer Center LAO
Locations (1):
- Yale University Cancer Center LAO, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm